CLINICAL TRIAL: NCT05830643
Title: Enhancing Consensual Social Skills to Prevent Non-consensual Sexual Acts: A Randomized Control Trial on Individuals With Problematic Sexual Interests in Children
Brief Title: Enhancing Consensual Social Skills to Prevent Non-consensual Sexual Acts
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022022
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2023-11

CONDITIONS: Paraphilias and Paraphilic Disorders
Keywords: Paraphilias; Pedophilia; Phallometry; Group psychotherapy; Social skills; Sexual arousal; Consent
MeSH Terms: conditions — Paraphilic Disorders; Pedophilia; Social Skills | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Intervention group (social skills focused psychotherapy) and control group (adult interest focused psychotherapy)
Who Masked: Outcomes Assessor
Masking Description: A Prospective Randomized Open, Blinded End-point (PROBE) design will occur. The end-points are evaluated by a blinded end-point clinical coordinator therefore there should be no different between the two types of trials in this regard.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social skills group psychotherapy (Experimental): Originally designed to meet the needs of patients with ASD or ASPD, this group is now popular with patients who want to work on issues involving their relationships with their probation or parole officers or in establishing health romantic relationships.
  Interventions: Behavioral: Social skills group psychotherapy
- Adult interest group psychotherapy (Active Comparator): The adult interest group has dual aims to (1) stop illegal sex acts and (2) enhance noncriminal sexual interests. The group focuses on respect for informed, voluntary, revocable, consent by examining various cognitive distortions that group members may endorse.
  Interventions: Behavioral: Adult interest group psychotherapy

INTERVENTIONS:
Behavioral: Social skills group psychotherapy — Groups are 1.5-hours and facilitated by a psychiatrist and social worker. The groups follow Cognitive Behavioral Therapy (CBT) and the Good Lives Model (GLM). Groups involve a check-in to receive advice from group members and then revolve around 1-2 topics. The facilitators are responsible for asking probing questions about the topic to facilitate group discussion and learning.
  CBT treatment involves efforts to change thinking patterns which might include: Learning to recognize one's distortions in thinking that are creating problems, and then to re-evaluate them. Gaining a better understanding of the behavior and motivation of others. Using problem-solving skills to cope with difficult situations.
  GLM conceptualized healthy sexuality as the natural outcome of success in achieving life goals. Some patients have difficulty changing their self-identity from that of "sex offender" to that of "former sex-offender". The GLM principles are helpful in achieving this aim.
  Other Names: Cognitive Behavioral Therapy (CBT); Good Lives Model (GLM)
  Arms: Social skills group psychotherapy
Behavioral: Adult interest group psychotherapy — Groups are 1.5-hours and facilitated by a psychiatrist and social worker. The groups follow Cognitive Behavioral Therapy (CBT) and the Good Lives Model (GLM). Groups involve a check-in to receive advice from group members and then revolve around 1-2 topics. The facilitators are responsible for asking probing questions about the topic to facilitate group discussion and learning.
  CBT treatment involves efforts to change thinking patterns which might include: Learning to recognize one's distortions in thinking that are creating problems, and then to re-evaluate them. Gaining a better understanding of the behavior and motivation of others. Using problem-solving skills to cope with difficult situations.
  GLM conceptualized healthy sexuality as the natural outcome of success in achieving life goals. Some patients have difficulty changing their self-identity from that of "sex offender" to that of "former sex-offender". The GLM principles are helpful in achieving this aim.
  Other Names: Cognitive Behavioral Therapy (CBT); Good Lives Model (GLM)
  Arms: Adult interest group psychotherapy

SUMMARY:
A challenge to Canadian society is the establishment of effective evidence-based interventions to prevent non-consensual sex acts. The Sexual Behaviours Clinic (SBC), located in Ottawa, Ontario, Canada, is an innovative and effective program devoted to the management of adults with persistent problematic sexual interests and behaviours (paraphilias). The primary aim of this project is to test the hypothesis that the SBC's success is due in part to its focus on consent and the enhancement of lawful and fulfilling social relationships (social skills). The study participants will include 60 voluntary male participants who have undergone an intake assessment with the SBC and show signs of paraphilic interests in children (based on the standard SBC intake questionnaire) who will be randomized into a social skills group or a control group focused on adult interests. Participants will attend these groups weekly for 3-months (12-weeks). Outcome measures will include pre-and-post social skills, sexual consent, sexual fantasy, and sexual urges surveys, pre-and-post phallometric testing (to test for objective sexual arousal), qualitative interviews of the study participants, their friends, and family members, and records of recidivism (self-report). Groups will be inclusive of individuals from varying ethnicities, backgrounds, sexual orientations, and intellectual and developmental levels.

DETAILED DESCRIPTION:
60 voluntary participants who have undergone an intake assessment with the SBC and show signs of paraphilic interests in children will be randomized into a control group or a social skills group. These groups have been running for ~15 years and the methods have been published (e.g., Fedoroff, 2020). A trained social worker and psychiatrist will facilitate the groups. Those in the control group will participate in a weekly group on adult interests for 3 months (12-weeks) and will receive the necessary psychological and/or pharmacological treatments needed for their condition. The intervention group will participate in a weekly group on consensual social skills for 3 months (12-weeks) and will receive the necessary psychological and/or pharmacological treatments needed for their condition. The groups will be compared in terms of any psychological or pharmacological treatments offered and received. It should be noted that the SBC has never offered treatment for homosexuality and does not propose to do so in this study.

Socio-demographic information of participants will be collected from a self-report measure completed at the participant's initial assessment, which is reviewed by the clinical coordinator. This questionnaire has been used in other studies completed within the SBC in the past. Participants will undergo phallometric testing to test for objective sexual arousal pre-and-post intervention. The clinical coordinator conducting the phallometric testing will be blinded to what group the participants are in. All participants will also complete baseline-standardized questionnaires including the Social Skills Inventory (SSI; Riggio, 1992), the revised Sexual Consent Scale (Humphreys & Brousseau, 2010), the Sexual Symptom Assessment Scale (SASS; Raymond et al., 2007), and the Fantasy Checklist (Bradford & Curry, 1991). They will complete the same questionnaires after attending the groups weekly for 3 months. In addition, after 3 months of Social Skills Therapy, a random group of 10 participants from the Social Skills group who have an identified significant other will be invited to participate in a semi-structured interview by a trained research assistant according to established qualitative methodology to investigate the efficacy of social skills therapy. Interviews will last 60-90 minutes, and a limited set of qualitative probes will revolve around the three broad themes explored during the quantitative portion of the study, namely, social skills, consent, and sexual interest. Boyatzis' (1998) principles of thematic analysis for data management and analysis will be used to analyze the overarching themes of the program. Whenever possible, analysis will be performed after each interview to inform the subsequent one, and to search for data saturation-defined as the time when no new information emerged from the interviews. Social skills and consent rubrics will structure the data analysis and coding process. An inductive process will be followed to add a quantitative understanding of the phenomenon under study.

ELIGIBILITY:
Inclusion Criteria:

* Male (sex at birth)
* 18 years of age or older
* Understand English
* Been assessed for a question of sexual interest in children

Exclusion Criteria:

* Cannot understand and/or read English
* Under the age of 18
* Does not have a penis
* Current or past history of psychoses
* In custody at the time of SBC assessment
* Participant shows no sexual interest in children
* Participant has already undergone group psychotherapy at the Sexual Behaviours Clinic

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Considering that a requirement for phallometric testing (which is the primary outcome tool used in the proposed study) is for the participant to have a penis, biological women will be excluded from this study. This does not include biological men who present their gender identity as female. While there is a test of objective sexual arousal designed for biological women (i.e., vaginal photoplethysmography, VPP), this method of measurement will not be used in the following study due to issues of validity with this measurement tool, as well as the difficulty in comparing the two methods of measurement. We recognize that women and adolescents of both genders also commit sex offences, however, in this study we plan to focus on the segment of the population at most risk of offending, adult males.
Enrollment: 60 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Penile Plethysmography/Phallometric Testing (PPG) | Approximately 2.5 hours to complete, depending on the length of time needed to return to baseline levels of arousal
  Objective measure of sexual arousal. Phallometry involves the physiological measurement of penile tumescence (i.e., erection) in response to various stimuli, such as audio descriptions of child and adult sexual interactions or pictures of nude or semi-clothed children and adults.

SECONDARY OUTCOMES:
Social Skills Inventory (SSI) | Approximately 10 minutes
  The brief Social Skills Inventory (SSI), also known as the Self-Description Inventory, is a 30-item Likert questionnaire that assesses 6 basic social skills that underlie social competence. It evaluates verbal (social) and non-verbal (emotional) communication skills and identifies strengths and weaknesses. As such, the SSI acts as a reliable and valid abilities measure of Emotional Intelligence.
Revised Sexual Consent Scale (SCS-R) | Approximately 10-20 minutes
  The Sexual Consent Scale-Revised (SCS-R) measures an individual's beliefs, attitudes, and behaviors with respect to how sexual consent should be and is negotiated between sexual partners. The SCS-R is a 39-item, Likert-type measure assessing both attitudes and behaviors with respect to sexual consent.
Sexual Symptom Assessment Scale (S-SAS) | Approximately 5-10 minutes
  In order to measure the severity of symptoms of Compulsive Sexual Behavior (CSB) the Sexual Symptom Assessment Scale (S-SAS) was developed. The S-SAS is a 12-item, self-rated scale, with each item scored 0-8; higher scores indicate more severe symptoms.
Fantasy Checklist | Approximately 10-20 minutes
  The fantasy checklist measures individual sexual fantasy using a 39-item, Likert scale with each item scored 0-6. Eight main factors corresponding to clearly identifiable fantasy themes have been identified (see Bradford, Curry, & Pawlak, 1996).

OTHER OUTCOMES:
Sociodemographic questionnaire | Approximately 30 minutes
  Socio-demographic information of participants will be collected from a self-report measure completed at the participant's initial assessment (Sexual Behaviours Clinic intake questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: John Bradford, MD, Principal Investigator — The Royal Ottawa Health Care Group (ROHCG); Dave Holmes, PhD, Principal Investigator — The Royal Ottawa Health Care Group (ROHCG); Emily Tippins, MSc, Study Director — The Royal Ottawa Health Care Group (ROHCG)
Locations (1):
- The Royal Ottawa Health Care Group (ROHCG), Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All applicable data will be shared on Mendeley Data once completed. Mendeley Data is a secure online repository for research data, permitting archiving of any file type and assigning a permanent and unique digital object identifier (DOI) so that the files can be easily referenced.
Supporting Information: Study Protocol, ICF
Time Frame: Starting February 2024.